CLINICAL TRIAL: NCT05775640
Title: PhD(c), RN, Lecturer
Brief Title: The Effect of Serious Game on Hospitalized Children's Anxiety, Fear, Knowledge, and Anxiety Levels in Their Parents
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Hilal PARLAK SERT, lecturer, Pamukkale University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: pau-parlaksert-001
Record Dates: First submitted 2023-02-23; First posted 2023-03-20 (Actual); Last update posted 2023-03-20 (Actual); Status verified 2023-03

CONDITIONS: Serious Game on Hospitalized Children
Keywords: Serious Game; Anxiety; Fear; Hospitalized Children; Parent
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Single blind pre-post test randomized controlled design
Who Masked: Participant
Masking Description: 32 control +32 intervention group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention): Sociodemographic data collection form, Clinical Information Form, The child medical fears scale, State and Trait Anxiety Inventory for Children were administered to the children in the control group, and the State-Trait Anxiety Inventory (STAI) was administered to the parents of the children in the control group on the 0th day of hospitalization. The standard clinical hospitalization process was not interfered with. On the third day of hospitalization, the children in the control group were administered the Clinical Information Form, the The child medical fears scale, the State and Trait Anxiety Inventory for Children, and the State-Trait Anxiety Inventory (STAI) for their parents. After the study, the link of the game was sent to the control group so that they could play the game in order to avoid ethical problems.
- intervention group (Experimental)
  Interventions: Behavioral: serious game

INTERVENTIONS:
Behavioral: serious game — The forms were applied to the children in the experimental group and the parents of the children on the 0th day of hospitalization. After the forms were applied, a serious game developed by the researchers was played. Children were given access to the game by giving a game link. The game can be played on digital platforms such as computers, tablets, etc. For children who do not have an electronic device, the game was downloaded to the computer in the hospital and the children were allowed to play. On the third day of hospitalization, the children and their parents were surveyed again and the Game Evaluation Questionnaire was filled. Access to the game will be closed at the end of the study.
  Arms: intervention group

SUMMARY:
Children may view hospitalization as a stressful experience. Children who are hospitalized show high levels of anxiety symptoms. During the hospitalization process, the family of the child as well as the children experience anxiety and stress. These fears and concerns are based on inadequate preparation for hospitalization and lack of knowledge.

Interventions to reduce the fear and anxiety of children during hospitalization include classical methods such as developing booklets and drawing pictures. While various benefits of these methods have been demonstrated, computer and web-based interventions have been shown to be the best way to prepare children for hospitalization. When computer and web-based interventions are examined, it is seen that they mostly focus on anxiety and pain control in children who are hospitalized for the operation process. More studies are needed to prepare hospitalized children for clinical procedures, to introduce the hospital environment, and to introduce the tools used in the hospital with computer and web-based interventions.

The research is a randomized controlled experimental study consisting of three stages. In the first stage of the research, serious game was developed. In the second stage, a randomized controlled study with experimental control group design was carried out. In the third stage, children's views and perceptions about serious play were determined and the effectiveness of the game was evaluated. The population of the research consisted of children aged 8-12, hospitalized in Pamukkale University Hospitals Pediatrics Service between October 2022 and February 2023. The G. Power program was used in the sample calculation and the sample size was calculated as 53 (Effect size 0.50, Power 95%). Considering that there may be data loss while collecting the data, it was increased by 20% and the experimental group was determined as 32 and the control group as 32.

ELIGIBILITY:
Inclusion Criteria:

* accept to participate in the study
* children hospitalized for the first time
* Inpatient treatment between the ages of 8-12-
* Comprehension and speech impairment
* without any mental disability
* Children and parents whose hospitalization is planned for at least three days

Exclusion Criteria:

* Daily and hospitalizations less than three days
* Repeated hospitalizations
* Speech, comprehension and mental problems
* Being treated for an oncological problem
* applied for trauma
* Children and parents who did not agree to participate in the study

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 64 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2022-10-26 (Actual); Study Completion 2023-03-30 (Estimated)

PRIMARY OUTCOMES:
Sociodemographic data collection form | applied on the first day of study
  It was developed the sociodemographic characteristics of the children and parents participating in the study
Clinical Information Form | up to 3 days
  includes information about the procedures, procedures, equipment and healthcare professionals used in the clinic.The form developed by the researchers includes information about the procedures, procedures, equipment and healthcare professionals used in the clinic. It consists of multiple-choice and 3-option questions.
The child medical fears scale | up to 3 days
  It is a scale to measure children's fears about medical procedures and practices.The total number of questions of the scale is 29, the lowest score obtained from the scale is 29, and the highest score is 87. The scale is a Likert type scale with three choices. Those who scored (0-29) on the scale were never afraid; (29-58) points are
State-Trait Anxiety Inventory for Children (STAI-CH) | up to 3 days
  It is used to measure the level of state and trait anxiety in children aged 9-12 who have reached literacy level.It aims to measure persistent individual differences as well as anxiety propensity. There are 20 items in total in the scale. The lowest score that can be obtained is 20, and the highest score is 60. Evaluates how the child usually feels according to the
State-Trait Anxiety Inventory for Adults(STAI) | up to 3 days
  It is one of the methods used to evaluate the level of anxiety.It consists of two subscales of 20 questions about state and trait anxiety. All questions are in a four-point Likert type. The scores of both subscales are summed separately and a total score between 20 and 80 is obtained. Higher scores indicate a higher
Game Evaluation Questionnaire | up to 3 days
  The developed game is prepared for children's evaluation.The questionnaire was developed in line with the literature. The survey consists of 2 parts. In the first part, the usefulness of the game is evaluated, and in the second part, the game content is evaluated.

CONTACTS AND LOCATIONS:
Locations (1):
- Pamukkale Universitesi, Denizli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No